CLINICAL TRIAL: NCT01599754
Title: Adjuvant Axitinib Treatment of Renal Cancer: A Randomized Double-blind Phase 3 Study of Adjuvant Axitinib vs. Placebo in Subjects at High Risk of Recurrent RCC
Brief Title: Adjuvant Axitinib Therapy of Renal Cell Cancer in High Risk Patients
Acronym: ATLAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary endpoint did not reach statistical significance
Sponsor: SFJ Pharma Ltd. II (Industry)
Collaborators: Pfizer (Industry); SFJ Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: SFJ Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AP311736
Record Dates: First submitted 2012-05-11; First posted 2012-05-16 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Clear Cell Renal Carcinoma
Keywords: renal cell carcinoma; axitinib; tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Axitinib (Experimental)
  Interventions: Drug: Axitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Axitinib — Axitinib 5 mg twice daily
  Other Names: Inlyta
  Arms: Axitinib
Drug: Placebo — Placebo twice daily
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine if adjuvant therapy with axitinib will prevent or delay the recurrence of renal cell cancer after surgery to remove the primary tumor in high risk patients.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind placebo controlled Phase 3 trial of oral axitinib starting at 5 mg twice daily given 3 years vs. placebo.

Approximately 700 patients will be randomized in a 1:1 ratio between axitinib vs placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients must be treated by nephrectomy and patients must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Patients must have no evidence of macroscopic residual disease or metastatic disease.
2. Male or female, age >=18 years (age >=20 years in Japan, Korea and Taiwan).
3. Patients must be diagnosed with one of the following based on American Joint Committee on Cancer (AJCC) TNM staging version 2010, Eastern Collaborative Oncology Group (ECOG) performance status (PS):

   * pT2, pN0 or pNx, M0 and ECOG PS 0-1
   * pT3, pN0 or pNx, M0 and ECOG PS 0-1
   * pT4, pN0 or pNx, M0 and ECOG PS 0-1
   * Any pT, pN1, M0 and ECOG PS 0-1
4. Patients must have histologically confirmed preponderant, defined as >50%, clear cell RCC.
5. Patients must not have received any previous systemic (includes chemotherapeutic, hormonal, or immunotherapeutic) treatment for RCC.
6. Patients must not have received any previous anti angiogenic treatment.
7. Patients must have adequate organ function.

Exclusion Criteria

1. Histologically undifferentiated carcinomas, sarcomas, collecting duct carcinoma, lymphoma, or patients with any metastatic renal sites.
2. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 hemorrhage <4 weeks of date of randomization.
3. Diagnosis of any non-RCC malignancy within the 5 years from date of randomization, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma of the cervix uteri that has been adequately treated with no evidence of recurrent disease for 12 months.
4. Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism.
5. Gastrointestinal abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2012-04; Primary Completion 2017-10-10 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (105):
- United States (25):
  - La Jolla, California
  - Los Angeles, California
  - Palo Alto, California
  - Pleasant Hill, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Ocala, Florida
  - Atlanta, Georgia
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Saint Paul, Minnesota
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - Albany, New York
  - New York, New York
  - Portland, Oregon
  - Charleston, South Carolina
  - Chattanooga, Tennessee
  - Austin, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Seattle, Washington
- China (12):
  - Beijing
  - Changchun
  - Chongqing
  - Dalian
  - Guangzhou
  - Hangzhou
  - Jinan
  - Nanchang
  - Shanghai
  - Suzhou
  - Tianjin
  - Wuhan
- France (11):
  - Besançon
  - Bordeaux
  - Hyères
  - Le Mans
  - Lyon
  - Marseille
  - Paris
  - Rennes
  - Saint-Herblain
  - Suresnes
  - Vandœuvre-lès-Nancy
- Hong Kong, Hong Kong
- India (18):
  - Ahmeadbad
  - Aurangabad
  - Bangalore
  - Chennai
  - Hyderabad
  - Karamsad
  - Kochi
  - Kolkota
  - Lucknow
  - Ludhiana
  - Mangalore
  - Manipal
  - Mumbai
  - Nashik
  - New Delhi
  - Pune
  - Surat
  - Visakhapatnam
- Japan (20):
  - Aichi
  - Akita
  - Aomori
  - Chiba
  - Fukuoka
  - Gifu
  - Hokkaido
  - Hyōgo
  - Kagawa
  - Kanagawa
  - Kumamoto
  - Kyoto
  - Nagasaki
  - Nigata-honmachi
  - Osaka
  - Shizuoka
  - Tokushima
  - Tokyo
  - Yamagata
  - Yamaguchi
- South Korea (6):
  - Busan
  - Daegu
  - Daejeon
  - Gyeonggi-do
  - Jeonnam
  - Seoul
- Spain (9):
  - Barcelona
  - Donostia / San Sebastian
  - Leganés
  - Llobregat
  - Madrid
  - Oviedo
  - Seville
  - Valencia
  - Zaragoza
- Taiwan (3):
  - Taichung
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Gross-Goupil M, Kwon TG, Eto M, Ye D, Miyake H, Seo SI, Byun SS, Lee JL, Master V, Jin J, DeBenedetto R, Linke R, Casey M, Rosbrook B, Lechuga M, Valota O, Grande E, Quinn DI. Axitinib versus placebo as an adjuvant treatment of renal cell carcinoma: results from the phase III, randomized ATLAS trial. Ann Oncol. 2018 Dec 1;29(12):2371-2378. doi: 10.1093/annonc/mdy454. PMID 30346481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 128 study sites in 9 countries randomized 724 participants into this study.
Groups:
- Axitinib: Participants at high risk of recurrent renal cell carcinoma (RCC) received Axitinib 5 milligram (mg) twice a day, in cycles of 4 weeks, up to 3 years with a minimum treatment duration of 1 year unless relapse, the occurrence of secondary malignancy or death occurred prior to 1 year. Participants were followed up after every 6 months after end of treatment.
- Placebo: Participants at high risk of RCC received placebo matched to Axitinib twice a day in cycles of 4 weeks, up to 3 years with a minimum treatment duration of 1 year unless relapse, the occurrence of secondary malignancy or death occurred prior to 1 year. Participants were followed up after every 6 months after end of treatment.
Period: Overall Study
Arm/Group | Axitinib | Placebo
Started | 363 | 361
Treated | 360 | 360
Completed | 0 | 1
Not Completed | 363 | 360
Not completed — Anticancer therapy need not in protocol | 5 | 2
Not completed — Participant noncompliance | 4 | 4
Not completed — Lost to Follow-up | 13 | 6
Not completed — Death | 31 | 33
Not completed — Adverse Event | 3 | 2
Not completed — Investigator decision | 1 | 3
Not completed — Withdrawal by Subject | 24 | 25
Not completed — Study terminated by sponsor | 282 | 285

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants regardless of whether or not treatment was administered and based on randomized treatment assignment.
Groups:
- Axitinib: Participants at high risk of recurrent RCC received Axitinib 5 mg twice a day, in cycles of 4 weeks, up to 3 years with a minimum treatment duration of 1 year unless relapse, the occurrence of secondary malignancy or death occurred prior to 1 year. Participants were followed up after every 6 months after end of treatment. .
- Total: Total of all reporting groups
Arm/Group | Axitinib | Placebo | Total
Number analyzed (Participants) | 363 | 361 | 724
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 255 | 247 | 502
  >=65 years | 108 | 114 | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (10.80) | 58.1 (11.33) | 58.0 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 111 | 194
  Male | 280 | 250 | 530
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 264 | 267 | 531
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 91 | 90 | 181
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  South Korea | 87 | 88 | 175
  Hong Kong | 6 | 5 | 11
  United States | 50 | 47 | 97
  Japan | 81 | 79 | 160
  China | 63 | 65 | 128
  Taiwan | 18 | 19 | 37
  France | 23 | 23 | 46
  India | 7 | 8 | 15
  Spain | 28 | 27 | 55
BMI [Count of Participants; unit: Participants] — Categorization of participants on body mass index (BMI): Normal (18.5 less than or equal to [<=] BMI less than [<] 25), Overweight + Obese (BMI greater than or equal to [>=] 25), Overweight (25<=BMI<30), Obese (BMI>=30) and Underweight (BMI<18.5).
  Participants
    Normal Weight | 187 | 173 | 360
    Overweight + Obese | 165 | 175 | 340
    Overweight | 115 | 124 | 239
    Obese | 50 | 51 | 101
    Underweight | 7 | 12 | 19
    Missing | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) as Assessed by Blinded Independent Review Committee (IRC)
Description: DFS is defined as time interval from the date of randomization to first date of recurrence/relapse (distant or local recurrence of [RCC] or occurrence of a secondary malignancy {occurrence of a second primary cancer other than RCC} or death). For participants with no DFS event, DFS was censored at date of last scan prior to time of analyses. Participants alive who did not have post-baseline disease assessments, DFS was censored at randomization. Participants who received further anti-tumor therapy prior to recurrence or occurrence of a secondary malignancy or death, DFS was censored on date of last scan prior to taking anti-tumor medication. Participants who missed 2 or more consecutive tumor scans immediately followed by an event were censored at date of last objective tumor assessment prior to missing/not readable scan.
Time Frame: From randomization date up to first date of recurrence or the occurrence of a secondary malignancy or death (up to 5 years)
Population: ITT population included all randomized participants regardless of whether or not treatment was administered and based on randomized treatment assignment.
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Axitinib: Participants at high risk of recurrent RCC received Axitinib 5 mg twice a day, in cycles of 4 weeks, up to 3 years with a minimum treatment duration of 1 year unless relapse, the occurrence of secondary malignancy or death occurred prior to 1 year. Participants were followed up after every 6 months after end of treatment.
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 363 | 361
years | NA [4.1 to NA] — Median and upper limit of CI was not estimable due to low number of participants who had event. | NA [4.1 to NA] — Median and upper limit of CI was not estimable due to low number of participants who had event.
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Test type: Superiority; p = 0.3211, Log Rank; Hazard Ratio (HR) = 0.870, 95% CI 2-sided [0.660 to 1.147]

2. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from the date of randomization to the date of death due to any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive. Participants lacking data beyond randomization had their survival times censored at randomization.
Time Frame: From randomization date until death due to any cause (up to 5 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 363 | 361
years | NA [NA to NA] — Median, upper and lower limit of CI was not estimable due to low number of participants who had event. | NA [NA to NA] — Median, upper and lower limit of CI was not estimable due to low number of participants who had event.
Statistical Analysis 1: Comparison: Axitinib vs Placebo; Test type: Superiority; p = 0.9246, Log Rank; Hazard Ratio (HR) = 1.026, 95% CI 2-sided [0.600 to 1.756]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AE) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Population: As-Treated population included all participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 360 | 360
Participants
  AEs | 353 | 333
  SAEs | 75 | 54

4. Secondary Outcome: Number of Participants With Treatment-Emergent Treatment Related Adverse Events and Serious Adverse Events (SAEs)
Description: A treatment related AE is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event had a causal relationship with the treatment or usage. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness was judged by investigator. AEs included both serious and non-serious adverse events.
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 360 | 360
Participants
  Treatment Related AEs | 326 | 202
  Treatment Related SAEs | 27 | 9

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) By Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AE was assessed according to severity as: Grade 1 (mild AE), Grade 2 (moderate AE), Grade 3 (severe AE), Grade 4 (life-threatening consequences) and Grade 5 (death related to AE).
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 360 | 360
Participants
  Grade 1 | 23 | 69
  Grade 2 | 108 | 152
  Grade 3 | 208 | 103
  Grade 4 | 12 | 8
  Grade 5 | 2 | 1

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities By Maximum CTCAE Grade: Hematology
Description: Hematology parameters included anemia, hemoglobin increased, lymphocyte count increased, lymphocyte count decreased, neutrophil count decreased, platelet count decreased, and white blood cell count decreased. CTCAE grades: Grade 1 (mild AE), Grade 2 (moderate AE), Grade 3 (severe AE), Grade 4 (life-threatening consequences) and Grade 5 (death related to AE).
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Population: As-Treated population included all participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received. Here, "number analyzed" signifies number of participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 360 | 360
Participants
  Anemia: number analyzed (Participants) | 351 | 355
  Anemia: Grade 1 | 256 | 233
  Anemia: Grade 2 | 87 | 114
  Anemia: Grade 3 | 8 | 6
  Anemia: Grade 4 | 0 | 2
  Anemia: Grade 5 | 0 | 0
  Hemoglobin increased: number analyzed (Participants) | 351 | 355
  Hemoglobin increased: Grade 1 | 328 | 354
  Hemoglobin increased: Grade 2 | 23 | 1
  Hemoglobin increased: Grade 3 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0
  Hemoglobin increased: Grade 5 | 0 | 0
  Lymphocyte count decreased: number analyzed (Participants) | 351 | 355
  Lymphocyte count decreased: Grade 1 | 305 | 282
  Lymphocyte count decreased: Grade 2 | 26 | 39
  Lymphocyte count decreased: Grade 3 | 19 | 33
  Lymphocyte count decreased: Grade 4 | 1 | 1
  Lymphocyte count decreased: Grade 5 | 0 | 0
  Lymphocyte count increased: number analyzed (Participants) | 351 | 355
  Lymphocyte count increased: Grade 1 | 343 | 339
  Lymphocyte count increased: Grade 2 | 0 | 0
  Lymphocyte count increased: Grade 3 | 8 | 16
  Lymphocyte count increased: Grade 4 | 0 | 0
  Lymphocyte count increased: Grade 5 | 0 | 0
  Neutrophil count decreased: number analyzed (Participants) | 351 | 355
  Neutrophil count decreased: Grade 1 | 284 | 299
  Neutrophil count decreased: Grade 2 | 48 | 45
  Neutrophil count decreased: Grade 3 | 19 | 8
  Neutrophil count decreased: Grade 4 | 0 | 3
  Neutrophil count decreased: Grade 5 | 0 | 0
  Platelet count decreased: number analyzed (Participants) | 349 | 354
  Platelet count decreased: Grade 1 | 267 | 303
  Platelet count decreased: Grade 2 | 77 | 49
  Platelet count decreased: Grade 3 | 5 | 1
  Platelet count decreased: Grade 4 | 0 | 1
  Platelet count decreased: Grade 5 | 0 | 0
  White blood cell count decreased: number analyzed (Participants) | 351 | 355
  White blood cell count decreased: Grade 1 | 288 | 281
  White blood cell count decreased: Grade 2 | 55 | 67
  White blood cell count decreased: Grade 3 | 8 | 6
  White blood cell count decreased: Grade 4 | 0 | 1
  White blood cell count decreased: Grade 5 | 0 | 0

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities By Maximum CTCAE Grade: Chemistry
Description: Chemistry parameters included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatine phosphokinase increased, creatinine increased, hypoalbuminemia, hypercalcemia, hypocalcemia, hyperglycemia, hypoglycemia, hyperkalemia, hypokalemia, hypernatremia, hyponatremia. CTCAE grades: Grade 1 (mild AE), Grade 2 (moderate AE), Grade 3 (severe AE), Grade 4 (life-threatening consequences) and Grade 5 (death related to AE).
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 360 | 360
Participants
  Alanine aminotransferase increased: number analyzed (Participants) | 2 | 6
  Alanine aminotransferase increased: Grade 1 | 1 | 2
  Alanine aminotransferase increased: Grade 2 | 0 | 3
  Alanine aminotransferase increased: Grade 3 | 0 | 0
  Alanine aminotransferase increased: Grade 4 | 1 | 1
  Alanine aminotransferase increased: Grade 5 | 0 | 0
  Alkaline phosphatase increased,: number analyzed (Participants) | 351 | 355
  Alkaline phosphatase increased,: Grade 1 | 298 | 316
  Alkaline phosphatase increased,: Grade 2 | 53 | 37
  Alkaline phosphatase increased,: Grade 3 | 0 | 2
  Alkaline phosphatase increased,: Grade 4 | 0 | 0
  Alkaline phosphatase increased,: Grade 5 | 0 | 0
  Aspartate aminotransferase increased: number analyzed (Participants) | 3 | 6
  Aspartate aminotransferase increased: Grade 1 | 0 | 1
  Aspartate aminotransferase increased: Grade 2 | 2 | 1
  Aspartate aminotransferase increased: Grade 3 | 1 | 3
  Aspartate aminotransferase increased: Grade 4 | 0 | 1
  Aspartate aminotransferase increased: Grade 5 | 0 | 0
  Blood bilirubin increased: number analyzed (Participants) | 351 | 355
  Blood bilirubin increased: Grade 1 | 315 | 330
  Blood bilirubin increased: Grade 2 | 30 | 18
  Blood bilirubin increased: Grade 3 | 6 | 6
  Blood bilirubin increased: Grade 4 | 0 | 1
  Blood bilirubin increased: Grade 5 | 0 | 0
  Creatine phosphokinase increased: number analyzed (Participants) | 2 | 2
  Creatine phosphokinase increased: Grade 1 | 0 | 0
  Creatine phosphokinase increased: Grade 2 | 0 | 0
  Creatine phosphokinase increased: Grade 3 | 0 | 0
  Creatine phosphokinase increased: Grade 4 | 2 | 1
  Creatine phosphokinase increased: Grade 5 | 0 | 1
  Creatinine increased: number analyzed (Participants) | 351 | 355
  Creatinine increased: Grade 1 | 13 | 7
  Creatinine increased: Grade 2 | 274 | 301
  Creatinine increased: Grade 3 | 60 | 46
  Creatinine increased: Grade 4 | 3 | 0
  Creatinine increased: Grade 5 | 1 | 1
  Hypoalbuminemia: number analyzed (Participants) | 351 | 355
  Hypoalbuminemia: Grade 1 | 347 | 348
  Hypoalbuminemia: Grade 2 | 4 | 5
  Hypoalbuminemia: Grade 3 | 0 | 2
  Hypoalbuminemia: Grade 4 | 0 | 0
  Hypoalbuminemia: Grade 5 | 0 | 0
  Hypercalcemia: number analyzed (Participants) | 351 | 355
  Hypercalcemia: Grade 1 | 335 | 344
  Hypercalcemia: Grade 2 | 16 | 11
  Hypercalcemia: Grade 3 | 0 | 0
  Hypercalcemia: Grade 4 | 0 | 0
  Hypercalcemia: Grade 5 | 0 | 0
  Hypocalcemia: number analyzed (Participants) | 351 | 355
  Hypocalcemia: Grade 1 | 280 | 266
  Hypocalcemia: Grade 2 | 64 | 85
  Hypocalcemia: Grade 3 | 3 | 4
  Hypocalcemia: Grade 4 | 2 | 0
  Hypocalcemia: Grade 5 | 2 | 0
  Hyperglycemia: number analyzed (Participants) | 351 | 355
  Hyperglycemia: Grade 1 | 116 | 115
  Hyperglycemia: Grade 2 | 160 | 159
  Hyperglycemia: Grade 3 | 62 | 56
  Hyperglycemia: Grade 4 | 12 | 23
  Hyperglycemia: Grade 5 | 1 | 2
  Hypoglycemia: number analyzed (Participants) | 351 | 355
  Hypoglycemia: Grade 1 | 230 | 246
  Hypoglycemia: Grade 2 | 111 | 101
  Hypoglycemia: Grade 3 | 9 | 6
  Hypoglycemia: Grade 4 | 0 | 1
  Hypoglycemia: Grade 5 | 1 | 1
  Hyperkalemia: number analyzed (Participants) | 351 | 355
  Hyperkalemia: Grade 1 | 318 | 325
  Hyperkalemia: Grade 2 | 1 | 0
  Hyperkalemia: Grade 3 | 26 | 21
  Hyperkalemia: Grade 4 | 6 | 9
  Hyperkalemia: Grade 5 | 0 | 0
  Hypokalemia: number analyzed (Participants) | 351 | 355
  Hypokalemia: Grade 1 | 340 | 348
  Hypokalemia: Grade 2 | 9 | 7
  Hypokalemia: Grade 3 | 0 | 0
  Hypokalemia: Grade 4 | 2 | 0
  Hypokalemia: Grade 5 | 0 | 0
  Hypernatremia: number analyzed (Participants) | 351 | 355
  Hypernatremia: Grade 1 | 245 | 245
  Hypernatremia: Grade 2 | 96 | 94
  Hypernatremia: Grade 3 | 8 | 14
  Hypernatremia: Grade 4 | 2 | 2
  Hypernatremia: Grade 5 | 0 | 0
  Hyponatremia: number analyzed (Participants) | 351 | 355
  Hyponatremia: Grade 1 | 331 | 338
  Hyponatremia: Grade 2 | 13 | 11
  Hyponatremia: Grade 3 | 0 | 0
  Hyponatremia: Grade 4 | 7 | 5
  Hyponatremia: Grade 5 | 0 | 1

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Thyroid Function
Description: Number of participants with thyrotropin levels: <5 milli-international units per litre (mIU/L), >=5 to <10 mIU/L, >=10 mIU/L are reported.
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Population: As-Treated population included all participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 351 | 356
Participants
  <5 mIU/L | 160 | 308
  >=5 - <10 mIU/L | 105 | 37
  >=10 mIU/L | 86 | 11

9. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Urinalysis
Description: Number of participants with urine protein dipstick grading: negative/trace (5 to 20 milligram per deciliter [mg/dL]), 1+ (30 mg/dL]), 2+ (100 mg/dL), 3+ (300 mg/dL) and 4+ (more than 1000 mg/dL) are reported.
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib | Placebo
Number analyzed (Participants) | 351 | 355
Participants
  Negative/trace | 135 | 237
  1+ | 88 | 84
  2+ | 74 | 24
  3+ | 49 | 8
  4+ | 5 | 2

ADVERSE EVENTS:
Time Frame: From Day 1 up to 28 days after last dose (maximum duration of 3 years)
Description: Same event may appear as both an AE and SAE. However,what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. As-Treated population consists of all participants who received at least 1 dose of study medication with treatment assignments designated according to actual study treatment received.
Arm/Group | Axitinib | Placebo
All-Cause Mortality (participants affected / at risk) | 31/360 | 33/360
Serious Adverse Events (participants affected / at risk) | 75/360 | 54/360
Other Adverse Events (participants affected / at risk) | 353/360 | 332/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=360) | Placebo (N=360)
Acute Coronary Syndrome (Cardiac disorders) | 3 | 0
Acute Myocardial Infarction (Cardiac disorders) | 3 | 1
Angina Pectoris (Cardiac disorders) | 2 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Stress Cardiomyopathy (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal Polyp (Gastrointestinal disorders) | 0 | 1
Large Intestinal Stenosis (Gastrointestinal disorders) | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal Disorder (Gastrointestinal disorders) | 1 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 2 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Biliary Colic (Hepatobiliary disorders) | 1 | 0
Cholangitis Acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 5 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Livery Injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diarrhoea Infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0
Otitis Media Chronic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 2 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1
Snake Bite (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of the Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 2 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 2 | 1
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal Disorder (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 1
Variococele (Reproductive system and breast disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic Intramural Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Peripheral Artery Aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=360) | Placebo (N=360)
Hypothyroidism (Endocrine disorders) | 73 | 22
Abdominal Pain (Gastrointestinal disorders) | 25 | 17
Abdominal Pain Upper (Gastrointestinal disorders) | 25 | 10
Consitpation (Gastrointestinal disorders) | 24 | 23
Diarrhoea (Gastrointestinal disorders) | 168 | 52
Dyspepsia (Gastrointestinal disorders) | 22 | 10
Nausea (Gastrointestinal disorders) | 36 | 34
Stomatitis (Gastrointestinal disorders) | 46 | 9
Vomiting (Gastrointestinal disorders) | 20 | 16
Asthenia (General disorders) | 41 | 22
Fatigue (General disorders) | 75 | 44
Malaise (General disorders) | 19 | 10
Pyrexia (General disorders) | 13 | 19
Nasopharyngitis (Infections and infestations) | 57 | 62
Upper Respiratory Tract Infection (Infections and infestations) | 33 | 32
Alanine Aminotransferase Increased (Investigations) | 31 | 13
Aspartate Aminotransferase Increased (Investigations) | 28 | 11
Blood Creatinine Increased (Investigations) | 34 | 23
Blood Thyroid Stimulating Hormone Increased (Investigations) | 48 | 5
Weight Decreased (Investigations) | 25 | 5
Weight Increased (Investigations) | 18 | 35
Decreased Appetite (Metabolism and nutrition disorders) | 45 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 59 | 36
Back Pain (Musculoskeletal and connective tissue disorders) | 46 | 54
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 21 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 11
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 35 | 23
Dizziness (Nervous system disorders) | 42 | 34
Dysgeusia (Nervous system disorders) | 24 | 5
Headache (Nervous system disorders) | 48 | 40
Insomnia (Psychiatric disorders) | 20 | 18
Proteniurea (Renal and urinary disorders) | 84 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 28
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 149 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 20 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 20 | 11
Dry Skin (Skin and subcutaneous tissue disorders) | 25 | 14
Palmar-Plantar Ertythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 115 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 31
Rash (Skin and subcutaneous tissue disorders) | 46 | 15
Hypertension (Vascular disorders) | 231 | 91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT01599754/SAP_000.pdf
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT01599754/Prot_001.pdf